CLINICAL TRIAL: NCT00040040
Title: Double-Blind, Placebo-Controlled Assessment of Potential Interactions Between IV Methamphetamine and Oral Bupropion
Brief Title: Assessment of Potential Interactions Between Methamphetamine and Bupropion - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of California, Los Angeles (Other)
Allocation: Randomized | Masking: Double | Purpose: Diagnostic
Other Study IDs: NIDA-CTO-0010-1
Record Dates: First submitted 2002-06-18; First posted 2002-06-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2003-08

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
The purpose of this study is to assess potential interactions between intravenous (IV) methamphetamine and oral bupropion.

DETAILED DESCRIPTION:
This is a human laboratory clinical pharmacology study to assess potential interactions between IV methamphetamine challenge and treatment with oral sustained-release bupropion.

ELIGIBILITY:
Inclusion Criteria:

Please contact site director for more details.

Exclusion Criteria:

Please contact site director for more details.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2002-06; Study Completion 2003-09

PRIMARY OUTCOMES:
Psychological effects
BP, HR

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - UCLA Integrated Substance Abuse Program, Los Angeles, California
  - University of Texas Health Science Center, Houston, Texas